CLINICAL TRIAL: NCT00984438
Title: Phase I/II Trial for Patients With Recurrent Resectable Glioblastoma Multiforme Using Surgery With Implantable BCNU Polymer Followed by Post-operative Irinotecan and Bevacizumab
Brief Title: Surgery With Implantable Biodegradable Carmustine (BCNU) Wafer Followed by Chemo for Patients With Recurrent Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: University of Cincinnati (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08081101
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2013-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Carmustine; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCNU wafter followed by chemotherapy (Experimental): Surgical Implantable BCNU wafer followed by Chemotherapy with Irinotecan and Bevacizumab for up to one year
  Interventions: Drug: BCNU Wafer; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: BCNU Wafer — Implantable during surgical resection into the tumor bed
  Other Names: Gliadel Wafer
Drug: Irinotecan — IV every 2 weeks for up to one year
  Other Names: CPT-11
Drug: Bevacizumab — IV every 2 weeks for up to one year
  Other Names: Avastin

SUMMARY:
The purpose of this research study is to try and identify a more effective treatment plan to improve survival rates for patients with a recurrent Glioblastoma Multiforme (GBM) brain tumor that can be removed by brain surgery.

The study will record what effects (good and bad) the combination of surgery with chemotherapy wafers inserted in the spot where the patient's tumor was during your surgery and post-operative chemotherapy has on the patient and their survival rate over the next 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of GBM in the past with MRI findings compatible with disease recurrence. Multifocal disease is permitted.
* Must have had prior treatment with standard doses of Temodar
* KPS >50; ECOG <3
* Predicted life expectancy of > 3 months
* Study entry must be within 5 weeks of surgical resection

Exclusion Criteria:

* Prior exposure to VEGF inhibitors or Irinotecan
* Intracranial bleed as defined by CT or MRI less than 6 months prior to entry
* GI bleed less than 6 months prior to entry
* Uncontrolled concurrent illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess disease free survival | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Margie Gerena-Lewis, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States